CLINICAL TRIAL: NCT06194149
Title: Assessment and Treatment of Loiasis With Positive Microfilaremia
Acronym: LoPoMi
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC23_0402
Record Dates: First submitted 2023-12-08; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Loiasis With Positive Blood Microfilaremia
Keywords: Loiasis; Microfilariae; epidemiology; treatment; complication
MeSH Terms: conditions — Loiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Loiasis is a vector-borne filariasis endemic in the forested areas in Central Africa whose incidence and morbi-mortality are poorly understood. Estimated prevalence is around 10 millions cases for a population around 30 million people. Considered to be a benign pathology, it has recently been associated with excess mortality, mainly in cases with major microfilaremia (> 8000 mf/ml).

Transmission is related to a mostly diurnal vector from the Chrysops genus. Adult worms are located in skin and subcutaneous tissues of infected patients. Females worms produce microfilariae which join bloodstream. Infected patients are mainly asymptomatic. Nevertheless, adult worms migration can lead to transient oedema (" œdème de Calabar ") ; adult worm can also be observed during subcunjonctival migration. Hypereosinophilia is also frequently encountered. Microfilariae presence in the bloodstream is asymptomatic, even in individuals with major microfilaremia.

Treatment differs according to the initial microfilaremia. There are three drugs available : diethylcarbamazine (DEC) ; albendazole (ALB) and ivermectin (IVM) each with different macrofilaricidal and microfiliaricidal activities. Several treatment guidelines based on the initial microfilaremia and drug activities have been proposed, on the basis of limited data. DEC is suggested for patients with microfilaremia < 2000 mf/ml. Regarding patients with microfilaremia between 2000 and 8000 mf/ml, initial treatment with IVM followed by DEC is suggested. Regarding patients with microfilaremia between 8000 mf/ml and 30000 mf/ml, initial treatment with IVM or ALB followed by DEC is suggested. Regarding patients with microfilaremia > 30000 mf/ml, initial treatment with ALB or apheresis is suggested to reduce blood microfilaremia, followed by DEC. All these guidelines are associated with major adverse events, mainly life-threatening encephalopathies. These adverse events are mostly encountered in patients with major blood microfilaremia.

The objective is to describe clinical characteristics, the management and clinical and biological evolution of patients with loiasis and positive blood microfilaremia.

DETAILED DESCRIPTION:
The protocol is based on the inclusion of patients diagnosed with loiasis with at least one positive blood microfilaremia > 0mf/ml between the 01/01/2000 and the 12/31/2022. Other inclusion criteria are specified below, including the necessity that patients were treated with a clinical and/or biological assessment after the first treatment.

Patients are screened using data available in the parasitology laboratories in tertiary centers in France (list of participating centers in progress). Data are collected in an anonymous way without identifying informations not requiring patients individual information. A local investigator at each center will collect the data then forward it to the main investigator. No correspondence list will be kept.

The primary outcome is focused on clinical and biological evolution after treatment for patients with loiasis and positive blood microfilaremia. Secondary outcomes are focused on the description of adverse events, description of initial clinical and biological characteristics and the description of therapeutic management. All outcomes are specified below.

Collected data are as follows :

* Initial data : demographic data (age at diagnosis, gender, country of origin, endemic country visited, length of stay, underlying conditions (HIV, hypertension, renal failure, immunosuppressive therapy, neoplasia)) / clinical data (current or previous symptoms possibly related to loasis: subcunjunctival migration, calabar swelling, pruritus, arthralgias, other types of manifestations (splenic, headache), length of symptoms, time between onset of symptoms and travel to endemic country / biological data (blood microfilaremia, blood count data (hemoglobin, blood hypereosinophilia, leucocytes) prior to treatment, creatininemia, proteinuria).
* Treatment data : treatment used (IVM, ALB or DEC) with duration and dosage if available, number of courses, use of combinations or sequential treatments, outpatient or inpatient treatment.
* Adverse events data : presence and description of adverse events / in particular, adverse events expected with treatment used in loasis: neurological disorders, hepatic cytolysis, renal impairment / percentage of adverse events requiring treatment discontinuation
* Evolution data : clinical assessment (vital status at last visit, at 6 months after treatment and 1 year after treatment (proportion of patients alive, deceased, lost to follow-up); for deceased patients: cause of death ; clinical evolution at last visit, at 6 months after treatment and 1 year after treatment (proportion of patients with symptoms related to loiasis)) / Biological assessment (microbiological evolution at last visit, 6 months after treatment and 1 year after treatment (proportion of patients with persistent microfilaremia/negative microfilaremia; median microfilaremia; proportion of patients with eosinophilia ≥ 0.5 G/L/having eosinophilia < 0.5 G/L; median eosinophilia)).

For descriptive analysis, quantitative data will be expressed as median or mean when the distribution is normal, while qualitative data will be expressed as a percentage. For comparative analyses, a Student's t test or a Mann Whitney test in the case of a non-normal distribution will be used to analyze quantitative data. A Chi2 test or a Fischer test in the case of a non-normal distribution will be used to analyze qualitative data. Survival analysis will be studied using a Kaplan Maier method. Any difference with a P < 0.05 will be considered significant.

The study results will enable the investigators to better describe the prognosis of patients with loiasis and positive blood microfilaremia , which is crucial to offer them appropriate management.

ELIGIBILITY:
Inclusion Criteria:

* Patient managed in one of the participating centers between the 01/01/2000 and the 12/31/2022
* Loiasis diagnosis with at least one positive blood microfilaremia > 0mf/ml
* Patient treated against loiasis
* At least one clinical and/or biological assessment after the first treatment dose

Exclusion Criteria:

- Patients not fulfilling inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our cohort study is composed of patients diagnosed with loiasis with at least one positive blood microfilaremia > 0mf/ml. Patients are screened using data avalaible in the parasitology laboratories in our partcipating centers. Data are collected anonimously.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Description of clinical and biological evolution of treated patients with loiasis and positive blood microfilaremia | At six months after treatment ; one year after treatment
  Vital status
Description of clinical and biological evolution of treated patients with loiasis and positive blood microfilaremia | At six months after treatment ; one year after treatment
  Reason of death for deceased patients / Clinical assessment
Description of clinical and biological evolution of treated patients with loiasis and positive blood microfilaremia | At six months after treatment ; one year after treatment
  percentage of patients with symptoms related to loiasis/ Biological assessment
Description of clinical and biological evolution of treated patients with loiasis and positive blood microfilaremia | At six months after treatment ; one year after treatment
  percentage of patients with persistent positive microfilaremia / median microfilaremia
Description of clinical and biological evolution of treated patients with loiasis and positive blood microfilaremia | At six months after treatment ; one year after treatment
  percentage of patients with hypereosinophilia > 0,5 G/l ; median eosinophilia

SECONDARY OUTCOMES:
Description of adverse events after treatment in patients with loiasis and positive blood microfilaremia | one year after treatment
  presence of adverse events and especially major adverse events (encephalopathy, acute kidney injury, hepatic cytolysis)

REFERENCES:
- [Background] Chesnais CB, Takougang I, Paguele M, Pion SD, Boussinesq M. Excess mortality associated with loiasis: a retrospective population-based cohort study. Lancet Infect Dis. 2017 Jan;17(1):108-116. doi: 10.1016/S1473-3099(16)30405-4. Epub 2016 Oct 21. PMID 27777031
- [Background] Boussinesq M. Loiasis: new epidemiologic insights and proposed treatment strategy. J Travel Med. 2012 May-Jun;19(3):140-3. doi: 10.1111/j.1708-8305.2012.00605.x. No abstract available. PMID 22530819
- [Background] Veletzky L, Eberhardt KA, Hergeth J, Stelzl DR, Zoleko Manego R, Mombo-Ngoma G, Kreuzmair R, Burger G, Adegnika AA, Agnandji ST, Matsiegui PB, Boussinesq M, Mordmuller B, Ramharter M. Distinct loiasis infection states and associated clinical and hematological manifestations in patients from Gabon. PLoS Negl Trop Dis. 2022 Sep 19;16(9):e0010793. doi: 10.1371/journal.pntd.0010793. eCollection 2022 Sep. PMID 36121900
- [Background] Bouchaud O, Matheron S, Loarec A, Dupouy Camet J, Bouree P, Godineau N, Poilane I, Cailhol J, Caumes E. Imported loiasis in France: a retrospective analysis of 167 cases with comparison between sub-Saharan and non sub-Saharan African patients. BMC Infect Dis. 2020 Jan 20;20(1):63. doi: 10.1186/s12879-019-4740-6. PMID 31959110
- [Background] Gardon J, Gardon-Wendel N, Demanga-Ngangue, Kamgno J, Chippaux JP, Boussinesq M. Serious reactions after mass treatment of onchocerciasis with ivermectin in an area endemic for Loa loa infection. Lancet. 1997 Jul 5;350(9070):18-22. doi: 10.1016/S0140-6736(96)11094-1. PMID 9217715
- [Background] Garcia A, Abel L, Cot M, Ranque S, Richard P, Boussinesq M, Chippaux JP. Longitudinal survey of Loa loa filariasis in southern Cameroon: long-term stability and factors influencing individual microfilarial status. Am J Trop Med Hyg. 1995 Apr;52(4):370-5. doi: 10.4269/ajtmh.1995.52.370. PMID 7741181